CLINICAL TRIAL: NCT02661763
Title: Prevalence of Rheumatic Heart Disease in Zambian Schoolchildren: an Echocardiographic Screening Study Involving Task-shifting to General Radiographers
Brief Title: Rheumatic Heart Disease Study in Lusaka
Status: Completed | Type: Observational
Sponsor: University of Zambia (Other)
Collaborators: University of Cape Town (Other); Novartis (Industry)
Responsible Party: Principal Investigator, John Musuku, Consultant Paediatrician / Cardiologist, University of Zambia
Other Study IDs: UNZABREC 002-10-13
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatic Heart Disease
Keywords: Rheumatic heart disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Schoolchildren in Zambia: Schoolchildren in grades 7-12 in fifteen randomly selected schools in Lusaka area

SUMMARY:
This study will determine the prevalence of rheumatic heart disease (RHD) in Lusaka, Zambia through school-based screening methodology using ultraportable echocardiography and a recently validated, abridged screening protocol based on World Heart Federation criteria. Children that screen positive for RHD at schools will undergo confirmatory evaluation at University Teaching Hospital (UTH), Lusaka's main referral hospital.

DETAILED DESCRIPTION:
It has been estimated that RHD affects over 32 million people worldwide, with the vast majority of cases occurring in the developing world. RHD is the most common cardiovascular disease in children and young adults and is a major cause of death in children above the age of 5 in many parts of the developing world, particularly sub-Saharan Africa.

RHD results from repeated attacks of acute rheumatic fever (ARF). ARF is a systemic inflammatory disease occurring mainly in children, characterized by fever, painful joints, and heart, skin, and neurological manifestations. ARF is linked with preceding Group A streptococcal (GAS) throat infections, which, if left untreated, carry an estimated 2-3% risk of developing ARF.

The pathologic hallmark of RHD is classically a valvulitis that affects mostly the mitral and/or aortic valves. Inflammation of the myocardium and pericardium may exacerbate the effects of valvular insufficiency, resulting in congestive heart failure, stroke and other complications. Over time, severe disability or death can ensue, especially in developing countries where the management of RHD patients is challenging and surgical interventions are not readily available.

ARF and RHD are diseases of poverty, especially in countries with limited healthcare systems. GAS thrives in situations of over-crowding where poor nutrition and sanitation are common and where medical treatment for sore throat is not readily available. For these reasons, RHD is endemic in many parts of the developing world, particularly sub-Saharan Africa, while it almost disappeared from most parts of the developed world (except for indigenous populations in some countries). It should be noted that the initial decline of ARF/RHD in the US and Europe most likely was due to improved living conditions and hygiene (primordial prevention), since it predated the introduction of penicillin.

RHD is one of few truly preventable chronic diseases. Currently, many sub-Saharan African countries do not focus efforts on primary and secondary prevention due to lack of resources. The long-term goal of an ongoing effort in Zambia is to develop capability to provide effective primary and secondary prevention of RHD, with the ultimate goal of eliminating new cases.

Although RHD is associated with major morbidity and mortality in children and young adults, until recently few reliable estimates of the burden from this disease existed in sub-Saharan Africa. Population-based screening for RHD had been limited to clinical examination, which does not detect early RHD in which a heart murmur or other clinical signs of disease are absent (subclinical disease). Estimates of RHD prevalence based on clinical surveillance methods compared with screening echocardiography have been shown to result in gross underestimates (up to 10 fold).

With advances in portable ultrasonography and the development of international guidelines for echocardiographic diagnosis of RHD, population-based screening for subclinical RHD is now possible. Using this new approach, recent studies in countries with similar geographic and demographic profiles to Zambia showed that RHD prevalence in sub-Saharan Africa is much higher than previously thought; approximately 1-3% of schoolgoing children appear to have evidence of definite or borderline RHD.

In this study, the investigators will apply echocardiographic screening methods to determine the prevalence of RHD in a large population of Zambian school children. Data on the disease burden of RHD in Zambia will be used to inform the design and conduct of health programs to combat RHD.

The proposed study will involve a sample size of at least 1,024 students in grades 7-12 in fifteen randomly selected schools in Lusaka. Each student that meets inclusion criteria will undergo a focused history and physical examination and rapid echocardiographic screening. The fifteen schools involved in the study will be identified as a random sample from 119 currently operating primary and secondary schools in Lusaka using standard sampling methods. Approximately 60-80 students from each school will be screened. The screening will be conducted using an ultraportable ultrasound device and an abridged screening protocol that has been validated in a separate study by investigators at the University of Cape Town in South Africa. Children with suspected ARF or RHD will be followed up at UTH for an in-depth clinical examination and quantitative electrocardiogram. Children with definite or borderline RHD according to World Heart Federation Criteria will be offered secondary penicillin prophylaxis according to national guidelines in Zambia. Children with sore throat will be referred for evaluation and treatment with penicillin according to national guidelines for primary prevention of RHD at UTH or a local health clinic.

An additional feature of this study is the development of local technical expertise to conduct echocardiographic screening. This is necessary because few health workers in Lusaka are proficient in cardiac echocardiography. The feasibility of task-shifting echocardiographic screening to non-expert health workers has been demonstrated in similar settings. The investigators will therefore train radiography technicians who have little or no previous experience with echocardiography to conduct school-based screening.

Given that radiographers will be newly trained to conduct screening echocardiography, two mechanisms will be implemented to help ensure successful school screening: (1) international echocardiography technician experts will periodically accompany study staff during school screenings to support the work of local radiographers; and (2) all screening echocardiograms will be de-identified and reviewed remotely by a professional third-party echocardiographer who will report back on any echocardiograms that are determined to be read as falsely negative by the field team.

Most data that will be obtained for the study will be entered through mobile electronic devices (computer tablets) at the time of capture into a digital system ("eRegister") that will be developed specifically for the study. The system uses DiMagi's "CommCare" platform, which includes a customizable mobile health data collection application and an online portal, "CommCareHQ," for secure data viewing and reporting. All access to the CommCare platform including mobile submissions will be done over HTTPS (hypertext transfer protocol) and will be cryptographically secure. Mobile devices will be password-locked and accessible only by the study staff member to whom the device is allocated. Once data are submitted to the server they will be automatically erased from the mobile device. Echocardiograms will also be saved in the system; images and videos will be temporarily stored on the hard drive of the ultrasound device and then transferred to the eRegister.

ELIGIBILITY:
Inclusion Criteria:

* Schoolgoing children in Lusaka in grades 7-12 at one of the participating primary or secondary schools
* Written parental consent
* Written assent by children
* Present on the day of school screening

Exclusion Criteria:

* Children whose parents do not provide consent
* Children who do not provide assent
* Children with health problems (e.g., skin infection of the chest) that preclude performance of transthoracic echocardiography

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A population of approximately 1,024 schoolchildren drawn from 15 primary and secondary schools in Lusaka, Zambia, to be screened for RHD in order to determine prevalence of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of RHD in Lusaka schoolchildren | Cross-sectional; the screening period is anticipated to last 5 months

CONTACTS AND LOCATIONS:
Overall Officials: John Musuku, Doctor, Principal Investigator — University of Zambia / University Teaching Hospital
Locations (1):
- University Teaching Hosptial, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carapetis JR, Steer AC, Mulholland EK, Weber M. The global burden of group A streptococcal diseases. Lancet Infect Dis. 2005 Nov;5(11):685-94. doi: 10.1016/S1473-3099(05)70267-X. PMID 16253886
- [Background] Marijon E, Ou P, Celermajer DS, Ferreira B, Mocumbi AO, Jani D, Paquet C, Jacob S, Sidi D, Jouven X. Prevalence of rheumatic heart disease detected by echocardiographic screening. N Engl J Med. 2007 Aug 2;357(5):470-6. doi: 10.1056/NEJMoa065085. PMID 17671255
- [Background] Bhaya M, Panwar S, Beniwal R, Panwar RB. High prevalence of rheumatic heart disease detected by echocardiography in school children. Echocardiography. 2010 Apr;27(4):448-53. doi: 10.1111/j.1540-8175.2009.01055.x. Epub 2010 Mar 24. PMID 20345448
- [Background] DiSciascio G, Taranta A. Rheumatic fever in children. Am Heart J. 1980 May;99(5):635-58. doi: 10.1016/0002-8703(80)90739-5. No abstract available. PMID 6989222
- [Background] Remenyi B, Wilson N, Steer A, Ferreira B, Kado J, Kumar K, Lawrenson J, Maguire G, Marijon E, Mirabel M, Mocumbi AO, Mota C, Paar J, Saxena A, Scheel J, Stirling J, Viali S, Balekundri VI, Wheaton G, Zuhlke L, Carapetis J. World Heart Federation criteria for echocardiographic diagnosis of rheumatic heart disease--an evidence-based guideline. Nat Rev Cardiol. 2012 Feb 28;9(5):297-309. doi: 10.1038/nrcardio.2012.7. PMID 22371105
- [Background] Kumar R. Controlling rheumatic heart disease in developing countries. World Health Forum. 1995;16(1):47-51. PMID 7873024
- [Background] Robertson KA, Volmink JA, Mayosi BM. Lack of adherence to the national guidelines on the prevention of rheumatic fever. S Afr Med J. 2005 Jan;95(1):52-6. PMID 15762250
- [Background] Marijon E, Mirabel M, Celermajer DS, Jouven X. Rheumatic heart disease. Lancet. 2012 Mar 10;379(9819):953-964. doi: 10.1016/S0140-6736(11)61171-9. PMID 22405798
- [Background] Kaplan EL. T. Duckett Jones Memorial Lecture. Global assessment of rheumatic fever and rheumatic heart disease at the close of the century. Influences and dynamics of populations and pathogens: a failure to realize prevention? Circulation. 1993 Oct;88(4 Pt 1):1964-72. doi: 10.1161/01.cir.88.4.1964. No abstract available. PMID 8403347
- [Background] Beaton A, Okello E, Lwabi P, Mondo C, McCarter R, Sable C. Echocardiography screening for rheumatic heart disease in Ugandan schoolchildren. Circulation. 2012 Jun 26;125(25):3127-32. doi: 10.1161/CIRCULATIONAHA.112.092312. Epub 2012 May 24. PMID 22626741
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Zuhlke LJ, Engel ME, Nkepu S, Mayosi BM. Evaluation of a focussed protocol for hand-held echocardiography and computer-assisted auscultation in detecting latent rheumatic heart disease in scholars. Cardiol Young. 2016 Aug;26(6):1097-106. doi: 10.1017/S1047951115001857. Epub 2015 Oct 1. PMID 26423122
- [Background] Engelman D, Kado JH, Remenyi B, Colquhoun SM, Watson C, Rayasidamu SC, Steer AC. Teaching focused echocardiography for rheumatic heart disease screening. Ann Pediatr Cardiol. 2015 May-Aug;8(2):118-21. doi: 10.4103/0974-2069.157024. PMID 26085762
- [Background] Colquhoun SM, Carapetis JR, Kado JH, Reeves BM, Remenyi B, May W, Wilson NJ, Steer AC. Pilot study of nurse-led rheumatic heart disease echocardiography screening in Fiji--a novel approach in a resource-poor setting. Cardiol Young. 2013 Aug;23(4):546-52. doi: 10.1017/S1047951112001321. Epub 2012 Oct 8. PMID 23040535
- [Background] Shmueli H, Burstein Y, Sagy I, Perry ZH, Ilia R, Henkin Y, Shafat T, Liel-Cohen N, Kobal SL. Briefly trained medical students can effectively identify rheumatic mitral valve injury using a hand-carried ultrasound. Echocardiography. 2013 Jul;30(6):621-6. doi: 10.1111/echo.12122. Epub 2013 Jan 24. PMID 23347259
- [Background] Carapetis JR. The stark reality of rheumatic heart disease. Eur Heart J. 2015 May 7;36(18):1070-3. doi: 10.1093/eurheartj/ehu507. Epub 2015 Jan 12. No abstract available. PMID 25583760
- [Background] Beaton A, Lu JC, Aliku T, Dean P, Gaur L, Weinberg J, Godown J, Lwabi P, Mirembe G, Okello E, Reese A, Shrestha-Astudillo A, Bradley-Hewitt T, Scheel J, Webb C, McCarter R, Ensing G, Sable C. The utility of handheld echocardiography for early rheumatic heart disease diagnosis: a field study. Eur Heart J Cardiovasc Imaging. 2015 May;16(5):475-82. doi: 10.1093/ehjci/jeu296. Epub 2015 Jan 5. PMID 25564396
- [Background] Engel ME, Haileamlak A, Zuhlke L, Lemmer CE, Nkepu S, van de Wall M, Daniel W, Shung King M, Mayosi BM. Prevalence of rheumatic heart disease in 4720 asymptomatic scholars from South Africa and Ethiopia. Heart. 2015 Sep;101(17):1389-94. doi: 10.1136/heartjnl-2015-307444. Epub 2015 Jun 15. PMID 26076935
- [Derived] Musuku J, Engel ME, Musonda P, Lungu JC, Machila E, Schwaninger S, Mtaja A, Mulendele E, Kavindele D, Spector J, Tadmor B, Gutierrez MM, Van Dam J, Colin L, Long A, Fishman MC, Mayosi BM, Zuhlke LJ. Prevalence of rheumatic heart disease in Zambian school children. BMC Cardiovasc Disord. 2018 Jul 3;18(1):135. doi: 10.1186/s12872-018-0871-8. PMID 29969998